CLINICAL TRIAL: NCT04632888
Title: The Effect of Telephone Support for Breastfeeding Follow-up on Physiological Jaundice, Exclusive Breastfeeding in the First Six Months, Infantile Colic, Maternal Breastfeeding Self-efficacy, and Breastfeeding Success
Brief Title: The Effect of Telephone Support for Breastfeeding Follow-up on Infantile Colic and Maternal Breastfeeding Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5762-GOA
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Breastfeeding, Exclusive; Infantile Colic; Self Efficacy; Jaundice, Neonatal
MeSH Terms: conditions — Breast Feeding; Colic; Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, parallel trial design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group/Telephone support for breastfeeding follow-up (Experimental): Study group: The women in the study group will be provided with a video call every day for the first week after discharge from the hospital, to provide consultancy to the mother on the matters she needs and to be recorded in the Baby Monitoring Form. The general appearance of the baby, observation during sucking, jaundice, drowsiness, reluctance to suck will be observed. The consultancy will be provided to the mother on these issues.
  In the following weeks, the consultancy will continue to be given to the study group by making a video talk one week apart.
  The researcher's phone will be given to the mothers in both groups and the incoming calls and their content will be recorded.
  Interventions: Other: Telephone support for breastfeeding follow-up
- Control Group (No Intervention): Control Group: No additional attempt or routine call will be made to mothers in the control group. The researcher's phone will be given to the mothers in both groups and the incoming calls and their content will be recorded.
  The control group will be called to fill in the scales for monitoring purposes.

INTERVENTIONS:
Other: Telephone support for breastfeeding follow-up — The researcher, after the mother is discharged, by making a video call by phone every day for the first week, providing counseling to the mother on matters that she needs and recording it in the Baby Monitoring Form The researcher gives the mother a video
  Arms: Study group/Telephone support for breastfeeding follow-up

SUMMARY:
This study was planned to examine the effect of telephone support for breastfeeding follow-up on physiological jaundice, exclusive breastfeeding in the first six months, infantile colic, maternal breastfeeding self-efficacy, and breastfeeding success.

DETAILED DESCRIPTION:
Hypothesis; H1: Telephone support for breastfeeding follow-up affects the development of physiological jaundice.

H2: Telephone support for breastfeeding monitoring affects exclusive breastfeeding for the first six months.

H3: Telephone support for breastfeeding follow-up affects infantile colic. H4: Telephone support for breastfeeding follow-up affects maternal breastfeeding self-efficacy.

H5: Telephone support for breastfeeding follow-up affects breastfeeding success of mothers.

Social media communication is planned to be completed at the 36th or older gestational week, who will have her first or second birth.

Block randomization will be applied according to maternal age, the number of births, baby gender, and birth week. Age (3 groups) X number of births (2 groups) X baby gender (2 groups) X gestational week (2 groups) = 24 blocks

Through social media, women between the ages of 18-45, who will have their first or second birth at their 36th or older gestational week will be included in the study. The woman in the control and study groups will be given breastfeeding and baby care training with the help of the training booklet by video calling.

* A socio-demographic data collection form will be filled, and the LATCH Breastfeeding Diagnostic Scale will be applied to the woman in the control and study groups on the day the mother gives birth, by making a video call by phone during breastfeeding.
* The women in the study group will be provided with a video call every day for the first week after their discharge from the hospital, to provide consultancy to the mother on the matters she needs and to be recorded in the Baby Monitoring Form. The general appearance of the baby, observation during sucking, jaundice, drowsiness, reluctance to suck will be observed. The consultancy will be provided to the mother on these issues.
* No additional intervention or routine call will be made to mothers in the control group. The researcher's phone will be given to the mothers in both groups and the incoming calls and their content will be recorded.
* In the following weeks, the consultancy will continue to be given to the working group by making a video talk one week apart. The control group will be called to fill in the scales for monitoring purposes.

ELIGIBILITY:
Inclusion Criteria:

* Having / had a new birth between the ages of 18-45
* Having his 1st or 2nd birth
* Agreeing to participate in the study voluntarily and obtaining consent form
* Having given birth to a healthy baby above 36 weeks of gestation
* Planning to breastfeed
* The baby does not need intensive care and does not develop any postpartum complications
* The baby does not have a vision and hearing problem, does not have a disease that may prevent breastfeeding
* The baby does not have a physical and psychological deficit
* The baby does not have a disease or an anatomical problem that will prevent breastfeeding
* Mother's ability to continue monitoring on the phone and to have a phone that can provide monitoring and video chat.
* No blood incompatibility between mother and baby.

Exclusion Criteria:

* Refusal to participate in the study
* Failure to continue monitoring by phone
* Mother's illiteracy
* Development of pathological jaundice in the baby

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The mothers with babies
Enrollment: 70 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
breastfeeding success | until discharge from the hospital an average 2 week
  LATCH Breastfeeding Assesment Scale: It is a measurement tool developed to evaluate breastfeeding. It was created to diagnose breastfeeding, to identify problems, to determine training accordingly, to create a common language among health professionals and to be used in studies. This measurement tool consists of the English initials of five evaluation criteria. Each item is scored between 0-2 points. The highest score is 10.
Infantile Colic | until discharge from the hospital an average 24 week
  Infantile Colic Scale: It was developed to diagnose and evaluate colic. The validity and reliability study of the scale was done in Turkey. 12 Scale items are graded with Likert type scoring ranging from 1 to 6.
Maternal Breastfeeding Self-Efficacy | until discharge from the hospital an average 24 week
  Breastfeeding Self-Efficacy Scale-Short Form: It is a 33-item scale to evaluate breastfeeding self-efficacy levels of mothers. Later, a 14-item short form of the scale was developed in 2003. It is applied more easily and evaluates self-efficacy correctly. Breastfeeding Self-Efficacy Short Form Scale is a 5 point Likert type scale.
rate of physiological jaundice | until discharge from the hospital an average 2 week
  physiological parameter of jaundice
rate of exclusive breastfeeding | until discharge from the hospital an average 24 week
  exclusive breastfeeding for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Principal Investigator — RN, PhD, Assoc. Prof.
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aykan Z, Ozalp Gerceker G. The effect of telephone-assisted breastfeeding monitoring on physiological jaundice, exclusive breastfeeding in the first six months, development of colic, and breastfeeding self-efficacy: A randomized controlled trial. Infant Behav Dev. 2025 Mar;78:102023. doi: 10.1016/j.infbeh.2024.102023. Epub 2024 Dec 31. PMID 39742561